CLINICAL TRIAL: NCT03193983
Title: V-Y Flap Versus Occlusive Dressing in Treating Fingertip Injuries With Exposed Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Abdelnasser Abdelfatah Farghay, Assiut University , resident doctor at orthopedic and trauma department assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssiutUMAAFDD
Record Dates: First submitted 2017-05-26; First posted 2017-06-21 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Injury Arm
Keywords: occlusive dressing
MeSH Terms: conditions — Arm Injuries | interventions — Occlusive Dressings

STUDY DESIGN:
Intervention Model Description: two groups Surgical group will undergo surgical coverage of the fingertip defect by V-Y flap using the skin on the volar aspect of the same finger designed as V shaped then mobilized dorsally to cover the defect and stitches to be Y shaped. Stitches are removed after 2 weeks.
  Conservative group will undergo minimal trimming of the bone end and an occlusive dressing that is changed on a weekly basis till complete healing of the defect that occurs after 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flaps Coverage (Experimental): Surgical group will undergo surgical coverage of the fingertip defect by V-Y flap using the skin on the volar aspect of the same finger designed as V shaped then mobilized dorsally to cover the defect and stitches to be Y shaped. Stitches are removed after 2 weeks.
  Interventions: Procedure: Flaps Coverage
- Occlusive Dressing (Experimental): Conservative group will undergo minimal trimming of the bone end and an occlusive dressing that is changed on a weekly basis till complete healing of the defect that occurs after 6 weeks.
  Interventions: Procedure: Occlusive Dressing

INTERVENTIONS:
Procedure: Flaps Coverage — Surgical group will undergo surgical coverage of the fingertip defect by V-Y flap using the skin on the volar aspect of the same finger designed as V shaped then mobilized dorsally to cover the defect and stitches to be Y shaped. Stitches are removed after 2 weeks.
  Arms: Flaps Coverage
Procedure: Occlusive Dressing — Conservative group will undergo minimal trimming of the bone end and an occlusive dressing that is changed on a weekly basis till complete healing of the defect that occurs after 6 weeks.
  Arms: Occlusive Dressing

SUMMARY:
Fingertip is a complex structure that is responsible for the fine function of the fingers and the whole hand. A fingertip injury is any soft tissue, nail or bony injury distal to the insertions of the long flexor and extensor tendons of a finger .Fingertip injury is a serious condition that if untreated properly could lead to significant functional disability and disuse of the injured finger. Up to date, defining the best treatment option for this injury remains controversial. Hand surgeons are divided between proponents of flap coverage and conservative treatment, driven by beliefs, training programs and financial aspects. After recently reviewing the literature for the current best evidence and fundamentals of conservative treatment, Krauss and Lalandei in their recent review of the literature, pointed out to the necessity for implementing controlled trials to compare both ways of treatment.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy and the results of occlusive dressing in treating fingertip injuries in comparison to flaps with much concern to certain factors that are closely related to our locality including patient compliance for regular follow up , functional outcome , time to return to work and its socioeconomical impact and cosmetic results .

Surgical group will undergo surgical coverage of the fingertip defect by V-Y flap using the skin on the volar aspect of the same finger designed as V shaped then mobilized dorsally to cover the defect and stitches to be Y shaped. Stitches are removed after 2 weeks.

Conservative group will undergo minimal trimming of the bone end and an occlusive dressing that is changed on a weekly basis till complete healing of the defect that occurs after 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* a. Inclusion criteria:

  1. Age Adults 12 - 60 years
  2. Diagnosis of fingertip injury with exposed bone (Allen type 2, 3 or 4) in any finger.
  3. Informed consent obtained by the patient.

Exclusion Criteria:

* · Old or complicated fingertip injuries.

  * Non-exposed bone fingertip injury (Allen type1).
  * Patients with severe debilitating disease.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
quick DASH score | 6 months
  A questionnaire consisting of eleven items that test the functional recovery following upper limb injury

SECONDARY OUTCOMES:
The presence of nail deformity. | 6 months
  any nail deformity will be reported the most common is hook nail deformity and then the deformity wiil be classified according to the severity to mild moderate and severe
Pulp volume compared to the contralateral finger: on lateral X-ray | 6 months
  either no decrease in the pulp volume or decreased to less than the half compared to the contralateral finger or more than the half compared to the contralateral finger
presence of painful neuroma | 6 months
  absent or present if present either affect patient function or not
Sensory related outcome in the form of Two point discrimination test (Weber index) | 6 months
  measurement and classification of Two point discrimination can be done by Touch-Test 2-Point Discriminator which consists of two sturdy, rotating, plastic disks that are joined together.Rounded tips are spaced at standard testing intervals from 1 to 15 mm apart. A 20 and 25 mm spacing also are given. One disk setting tests from 1 to 8mm, and the other setting tests from 9 to 15 mm. To change settings, just rotate the top disk until it clicks in place
Finger length: expressed as a shortage in mm. compared to contralateral finger. | 6 months
  the shortage is classified to three items a) no shortage b) less half compared to contralateral finger and c) more than compared to contralateral finger

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
whole study data and results will be available